CLINICAL TRIAL: NCT02035644
Title: Study on the Efficacy aNd Safety of Jinlida Granules in Patients With Inadequately cOntrolled tYpe-2 Diabetes and dysLIpidemia Under liFe Style Intervention (ENJOY LIFE Study)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: Shijiazhuang Yiling Pharmaceutical Co. Ltd (Industry)
Responsible Party: Principal Investigator, Guang Ning, the vice-president of Shanghai Jiao Tong University Affiliated Ruijin Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CCEMD021
Record Dates: First submitted 2014-01-12; First posted 2014-01-14 (Estimated); Last update posted 2014-01-14 (Estimated); Status verified 2014-01

CONDITIONS: Type 2 Diabetes; Dyslipidemia
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Dyslipidemias

ARMS (2):
- Jinlida granules (Experimental): Jinlida granules, a traditional Chinese medicine, was a herbal formula which was developed under cognition of the theory in the onset of diabetes
  Interventions: Drug: Jinlida granules
- placebo granules (Placebo Comparator): placebo prepared in indistinguishable granules
  Interventions: Drug: placebo granules

INTERVENTIONS:
Drug: Jinlida granules
  Arms: Jinlida granules
Drug: placebo granules
  Arms: placebo granules

SUMMARY:
The aim of the present study is to evaluate the efficacy and safety of Jinlida granules in patients with inadequately controlled type-2 diabetes and dyslipidemia under life style intervention.

ELIGIBILITY:
Inclusion Criteria:

1. age of 20-70 years;
2. diagnosed with type 2 diabetes inadequately controlled under life style intervention with 3 months before screening;
3. HbA1c ≥6.5% and ≤10.0%, and fasting plasma glucose ≥7 and ≤13.3mmol/L at baseline;
4. diagnosed with dislipidemia with triglycerides>150mg/dL (1.70mmol/L), and/or total cholesterol >200mg/dL (5.16mmol/L), and/or LDL-c>100mg/dL (2.58mmol/L)
5. body mass index (BMI): 20<BMI<40 kg/m2;

Exclusion Criteria:

1. moderate or severe liver dysfunction, abnormal renal function;
2. severe dysfunction of the heart;
3. histories of acute diabetic complications including diabetic ketoacidosis or hyperosmolar hyperglycemic non-ketotic coma within 3 months;
4. psychiatric disease or severe infection;
5. pregnancy or planned pregnancy;
6. use of any drug (including insulin) for treatment of diabetes or dyslipidemia within 3 months;
7. use of chronic (>7 days) systemic glucocorticoid therapy within 8 weeks or receive growth hormone therapy within 6 months;
8. diagnosed with type 1 diabetes, or gestational diabetes, or other specific types of diabetes;
9. history of malignant tumor within 5 years.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2014-02; Primary Completion 2015-02 (Estimated)

PRIMARY OUTCOMES:
change in HbA1c levels | 16 weeks

SECONDARY OUTCOMES:
fasting, postload 30-min and 2-h plasma glucose | 16 weeks
fasting, postload 30-min and 2-h serum insulin | 16 weeks
serum lipids | 16 weeks
glucose disposal rate (GDR) values from hyperinsulinemic euglycemic clamp | 16 weeks
incretins | 16 weeks
metabolomic parameters | 16 weeks
BMI | 16 weeks
blood pressures | 16 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Guang Ning, Shanghai, Shanghai Municipality, China